CLINICAL TRIAL: NCT03677778
Title: Interscalene Brachial Plexus Block Washout to Reverse Inadvertent Phrenic Nerve Blockade
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Stanford University (Other)
Responsible Party: Principal Investigator, Chi-Ho Ban Tsui, Professor, Stanford University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 46830
Record Dates: First submitted 2018-09-18; First posted 2018-09-19 (Actual); Last update posted 2022-08-02 (Actual); Status verified 2022-07

CONDITIONS: Anesthesia, Local; Phrenic Nerve Paralysis; Upper Extremity Injury; Phrenic Nerve Palsy on the Left; Phrenic Nerve Palsy on the Right
MeSH Terms: conditions — Arm Injuries

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo group (Placebo Comparator): After surgery, in the post-operative recovery room, patients randomized to both the intervention and control groups will have 10cc 0.5% ropivacaine bolused via their nerve catheters. After 30 minutes, the following will be measured/assessed: spirometry data, pain scores (using the Numeric Rating Scale), and, if time is sufficient, bilateral diaphragmatic excursion via ultrasonography and brachial plexus motor and sensory exams. This control group will have no normal saline injected into their nerve catheter (no intervention). Then, both the control and treatment groups will have the following measured/assessed after 5, 15 and 30 minutes: spirometry data, pain scores (using the Numeric Rating Scale), and, if time is sufficient, bilateral diaphragmatic excursion via ultrasonography and brachial plexus motor and sensory exams. Investigators will be blinded to whether the patient is in the intervention or treatment group.
  Interventions: Other: Placebo
- Treatment group (Active Comparator): After surgery, in the post-operative recovery room, patients randomized to both the intervention and control groups will have 10cc 0.5% ropivacaine bolused via their nerve catheters. After 30 minutes, the following will be measured/assessed: spirometry data, pain scores (using the Numeric Rating Scale), and, if time is sufficient, bilateral diaphragmatic excursion via ultrasonography and brachial plexus motor and sensory exams. This group will then have 30ml of normal saline injected into their nerve catheter. Then, both the control and treatment groups will have the following measured/assessed after 5, 15 and 30 minutes: spirometry data, pain scores (using the Numeric Rating Scale), and, if time is sufficient, bilateral diaphragmatic excursion via ultrasonography and brachial plexus motor and sensory exams. Investigators will be blinded to whether the patient is in the intervention or treatment group.
  Interventions: Procedure: Normal saline injected via interscalene nerve catheter

INTERVENTIONS:
Procedure: Normal saline injected via interscalene nerve catheter — With the catheter covered, treatment group patients will receive a normal saline (NS) bolus regimen (30cc 0.9% NS) via their interscalene nerve block catheter.
  Arms: Treatment group
Other: Placebo — With the catheter covered, placebo group patients will go through the same steps as the treatment group, but no solution will be injected into the interscalene nerve block catheter.
  Arms: Placebo group

SUMMARY:
One of the most frequently performed peripheral nerve blocks (the injection of local anesthetic near nerves to block sensation/ movement to a specific part of the body) is the interscalene brachial plexus block for upper extremity surgeries. This type of block can unmask underlying respiratory issues such as shortness of breath due to a well-known and typically insignificant side effect of temporary diaphragmatic paralysis.

The nerve block may be able to use saline solution to wash out the local anesthetic and potentially reverse this respiratory side effect. Specifically, the goal of this study is to determine if the injection of saline through the nerve block catheter reverses blockade of the phrenic nerve supplying the diaphragm, without affecting the ability of the nerve block to provide pain control after surgery.

ELIGIBILITY:
Inclusion criteria:

* All adult patients (18 years and over) scheduled for surgery requiring a continuous interscalene brachial plexus nerve block catheter as part of their anesthetic care.

Exclusion criteria:

* Concomitant life-threatening injuries and other concomitant injuries causing significant pain
* Pregnant
* Any condition impairing patient's ability to consent to participation in study, and an existing condition contraindicating a nerve block, i.e. nerve injury, existing bleeding disorder, infection in the vicinity of the block, and patient refusal.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 43 (Actual)
Dates: Start 2018-10-22 (Actual); Primary Completion 2022-07-07 (Actual); Study Completion 2022-07-07 (Actual)

PRIMARY OUTCOMES:
Change in forced vital capacity (FVC) | Before the nerve block placement, within 1 hour after the surgery, then in 5, 15, and 30 minutes after the saline injection/placebo (1 minute each for a total of 5 assessments)
  Spirometry data will be collected using a digital spirometer before nerve block is placed, after surgery, and after receiving either the placebo or treatment.
Change in peak expiratory flow (PEF) | Before the nerve block placement, within 1 hour after the surgery, then in 5, 15, and 30 minutes after the saline injection/placebo (1 minute each for a total of 5 assessments)
  Spirometry data will be collected using a digital spirometer before nerve block is placed, after surgery, and after receiving either the placebo or treatment.
Change in forced expiratory volume in 1 second (FEV1) | Before the nerve block placement, within 1 hour after the surgery, then in 5, 15, and 30 minutes after the saline injection/placebo (1 minute each for a total of 5 assessments)
  Spirometry data will be collected using a digital spirometer before nerve block is placed, after surgery, and after receiving either the placebo or treatment.

SECONDARY OUTCOMES:
Diaphragmatic excursion | Before nerve block is placed, within 1 hour after the surgery, and while receiving either the placebo or treatment (5 minutes each for a total of 3 assessments.)
  Diaphragmatic excursion will be assessed via ultrasound before nerve block is placed, after surgery, and while receiving either the placebo or treatment.
Brachial plexus sensory and motor exam | Before nerve block is placed, within 1 hour after the surgery, and while receiving either the placebo or treatment (2 minutes each for a total of 3 assessments).
  Brachial plexus sensory and motor exam changes will be assessed before nerve block is placed, after surgery, and while receiving either the placebo or treatment.
Pain scores | Pain scores will be assessed before nerve block is placed, within 1 hour after the surgery, while receiving either the placebo or treatment. (1 minute each for a total of 3 assessments)
  The Numerical Pain Rating Scale is a subjective measure in which individuals rate their pain on an eleven-point numerical scale. The scale is composed of 0 (no pain at all) to 10 (worst imaginable pain). Pain scores will be assessed before nerve block is placed, after surgery, while receiving either the placebo or treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Ban Tsui, MD, Principal Investigator — Stanford University
Locations (1):
- Stanford Health Care (SHC), Palo Alto, California, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Urmey WF, Talts KH, Sharrock NE. One hundred percent incidence of hemidiaphragmatic paresis associated with interscalene brachial plexus anesthesia as diagnosed by ultrasonography. Anesth Analg. 1991 Apr;72(4):498-503. doi: 10.1213/00000539-199104000-00014. PMID 2006740
- [Background] Urmey WF, McDonald M. Hemidiaphragmatic paresis during interscalene brachial plexus block: effects on pulmonary function and chest wall mechanics. Anesth Analg. 1992 Mar;74(3):352-7. doi: 10.1213/00000539-199203000-00006. PMID 1539813
- [Background] Lenters TR, Davies J, Matsen FA 3rd. The types and severity of complications associated with interscalene brachial plexus block anesthesia: local and national evidence. J Shoulder Elbow Surg. 2007 Jul-Aug;16(4):379-87. doi: 10.1016/j.jse.2006.10.007. Epub 2007 Apr 19. PMID 17448698
- [Background] Zink W, Graf BM. Local anesthetic myotoxicity. Reg Anesth Pain Med. 2004 Jul-Aug;29(4):333-40. doi: 10.1016/j.rapm.2004.02.008. PMID 15305253
- [Background] Katircioglu K, Ozkalkanli MY, Kalfaoglu H, Sannav S, Ozgurbuz U, Savaci S. Reversal of prilocaine epidural anesthesia using epidural saline or ringer's lactate washout. Reg Anesth Pain Med. 2007 Sep-Oct;32(5):389-92. doi: 10.1016/j.rapm.2007.06.004. PMID 17961836
- [Background] Park EY, Kil HK, Park WS, Lee NH, Hong JY. Effect of epidural saline washout on regression of sensory and motor block after epidural anaesthesia with 2% lidocaine and fentanyl in elderly patients. Anaesthesia. 2009 Mar;64(3):273-6. doi: 10.1111/j.1365-2044.2008.05746.x. PMID 19302639
- [Background] Sitzman BT, DiFazio CA, Playfair PA, Stevens RA, Hanes CF, Herman TB, Yates HK, Leisure GS. Reversal of lidocaine with epinephrine epidural anesthesia using epidural saline washout. Reg Anesth Pain Med. 2001 May-Jun;26(3):246-51. doi: 10.1053/rapm.2001.22587. PMID 11359224
- [Background] Ip VH, Tsui BC. Continuous interscalene block: the good, the bad and the refined spread. Acta Anaesthesiol Scand. 2012 Apr;56(4):526-30. doi: 10.1111/j.1399-6576.2012.02650.x. Epub 2012 Feb 16. PMID 22338616
- [Background] Courtney KR, Kendig JJ, Cohen EN. Frequency-dependent conduction block: the role of nerve impulse pattern in local anesthetic potency. Anesthesiology. 1978 Feb;48(2):111-7. No abstract available. PMID 306789
- [Derived] Gerber LN, Sun LY, Ma W, Basireddy S, Guo N, Costouros J, Cheung E, Boublik J, Horn JL, Tsui BC. Clinical effect of normal saline injectate into interscalene nerve block catheters given within one hour of local anesthetic bolus on analgesia and hemidiaphragmatic paralysis. Reg Anesth Pain Med. 2021 Feb;46(2):124-129. doi: 10.1136/rapm-2020-101922. Epub 2020 Nov 12. PMID 33184166